CLINICAL TRIAL: NCT02271750
Title: A Study of Insulin-like Growth Factors and Other Neurotrophic Factors in the Cerebrospinal Fluid From Patients With Dementia
Brief Title: IGF and Other Neurotrophic Factors in Patients With Dementia
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Dementia IGF; 1-10-72-250-14 (Registry Identifier: The National Committee on Health Research Ethics (Denmark))
Record Dates: First submitted 2014-10-02; First posted 2014-10-22 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2014-10

CONDITIONS: Dementia
Keywords: IGF, Neurotrophic factors, Dementia, spinal fluid
MeSH Terms: conditions — Dementia | interventions — Spinal Puncture

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — spinal fluid and blood sample for identification of different factors
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dementia
  Interventions: Procedure: lumbar puncture
- controls
  Interventions: Procedure: lumbar puncture

INTERVENTIONS:
Procedure: lumbar puncture — for spinal fluid

SUMMARY:
The global prevalence of dementia is close to 36 million (2010). Furthermore the number is predicted to double in the next 20 years, primarily due to the demographic ageing. A perspective that will challenge the current healthcare systems and national economies.

Dementia is characterized by progressive deterioration in cognition, function and behavior that is sufficiently severe to compromise social and occupational functioning.

The pathogenesis of dementia remains elusive. Thus, there is a need to increase our understanding of the mechanisms leading to the most common forms of dementia. A better understanding of the disease may enable an earlier diagnosis and importantly, a causal treatment of Alzheimer as opposed to the merely symptomatic options available to day.

An experiment with rats and memory might already have taken the first step towards this. The experiment has demonstrated that administration of IGF-II to rats significantly enhances memory retention and prevents forgetting. Furthermore inhibitory avoidance learning leads to an increase in the hippocampal expression of IGF-II. Finally, yet importantly, injections of recombinant IGF-II into hippocampus after training or memory retrieval significantly enhance memory retention and prevent forgetting.

The spinal fluid and the serum will be analysed at the Medical Research Laboratory. The immunological concentrations of IGF-I and -II are measured by validated in-house analyses. Furthermore, Aarhus University Hospital has a unique technique, whereby it is possible to measure the bioactivity of IGF-I and -II in the cerebrospinal fluid. The concentrations of NGF, BDNF and sCD-163 in spinal fluid and serum will be analysed by already established techniques.

The purpose of this study is therefore to define the concentration and biological activity of IGF-I, IGF-II, BDNF, NGF and sCD-163 in the cerebrospinal fluid and serum in patients with Alzheimer's compared with controls.

DETAILED DESCRIPTION:
Introduction Dementia The estimated prevalence of dementia in Denmark is 85.000 (2011) and the global prevalence is close to 36 million (2010). Furthermore the number is predicted to double in the next 20 years, primarily due to the demographic ageing. The costs of dementia accounts for 1% of the world's GDP - a perspective that will challenge the current healthcare systems and national economies (1,2,3).

Dementia includes a number of progressive degenerative brain diseases. Dementia is characterized by progressive deterioration in cognition, function and behavior that is sufficiently severe to compromise social and occupational functioning. Dementia is characterized by loss of episodic memory, difficulty in naming and word finding, apraxia, executive dysfunction and changes in personality and mood. The most common cause of dementia is Alzheimer's disease (4, 5, 6).

The pathogenesis of Alzheimer dementia remains elusive. For many years the pathophysiological hallmark of Alzheimers dementia has been the toxicity caused by the accumulation of the proteins amyloid-beta in plaques and phosphorylated tau associated with neurofibrillary tangles. However, this theory is based on the genetic "early-onset familial Alzheimers", which is a less frequent inherited type. Currently, the hypotheses on the pathogenesis of Alzheimer actually disagree with that of the amyloid-beta theory. Thus, there is a need to increase our understanding of the mechanisms leading to the most common forms of Alzheimer's disease. A better understanding of the disease may enable an earlier diagnosis and importantly, a causal treatment of Alzheimer as opposed to the merely symptomatic options available to day (4, 7, 8, 9).

IGF-system One of the main areas of recent research in dementia is the role of neurotrophic support, a research area which embraces insulin and the insulin-like growth factor system. Insulin and the IGF system are important in normal somatic growth, development, tissue repair and regeneration throughout life. Earlier studies have indicated that impairments in cerebral glucose utilization and energy metabolism represent very early abnormalities that precede or accompany the initial stages of cognitive impairment. However, type 2 diabetes, which is often characterized by insulin resistance, has not been established as a cause of Alzheimer although there is a correlation between insulin resistance and cognitive dysfunction.

The cellular signaling pathways of IGF-I and IGF-II overlap to a great extent with the pathways used by insulin, and all three proteins bind to the same receptors though with different affinities. Several studies have shown that the ratio between the concentrations of IGF-I in cerebrospinal fluid (CSF) and plasma (the CSF/plasma ratio) is reduced in Alzheimer patients. Interestingly, IGF-I seems to promote amyloid-beta clearance.

IGF-II has been less studied but it is expressed in the brain both during development and in adulthood and declines with ageing. In the brain the relative concentration is highest in the hippocampus. (10-14). Furthermore, our group has novel data indicating that in CSF, IGF-II is the most important growth factor when it comes to activating the IGF-I receptor (Mia-Maiken Kallestrup et al., manuscript in preparation).

Memory Memory is a question of consolidation whereby newly learned labile information becomes stronger and resilient to disruption. This process depends on de novo RNA and protein synthesis and the function of the cAMP response element binding protein (CREB) and the CCAAT enhancer binding protein (C/EBP), both of which are transcription factors. Former studies have shown that there is a binding site for C/EBP in the promoter region of the IGF-II gene in liver and other tissues (10).

IGF-II and memory To solve the puzzle of dementia it is important to explain early changes in biomarkers in early stages of dementia and thereby possibly reveal the pathogenesis and possible treatments. An experiment with rats and memory might already have taken the first step towards this. It has been demonstrated that administration of IGF-II to rats significantly enhances memory retention and prevents forgetting. Furthermore inhibitory avoidance learning (a paradigm in which the subject learns to associate a particular context with the occurrence) leads to an increase in the hippocampal expression of IGF-II. Finally, yet importantly, injections of recombinant IGF-II into hippocampus after training or memory retrieval significantly enhance memory retention and prevent forgetting (10).

Neurotrophic growth factors:

The human adult brain is able to generate new neurons even though it has a limited capacity. Possibly this capacity depends on sufficient neurotrophic growth factors. The neurotrophic factors include nerve growth factor (NGF) and brain derived neurotrophic factor (BDNF).

BDNF is important in neuronal survival, synaptic plasticity and memory, which along with the tendency of increased levels of BDNF in early stages of Alzheimer's indicate a connection. The increase of BDNF in early stages of Alzheimer's could be a reflection of compensation for the neurodegeneration. During the progression of Alzheimer's the level of BDNF is decreasing to a level of healthy elderly people.

NGF induces growth of neurons and maintains neuron proliferation interacting with other growth factors. Levels of NGF in serum, CSF or brain do not seem to differ from Alzheimer's patients to normal elderly patients but seem to vary between different brain regions. Finally the expression pattern of BDNF and NGF highly correlates with amyloid concentration (15).

Cluster of differentiation 163(CD-163) CD-163 is a scavenger receptor, which recognizes and uptakes macromolecules for the hemoglobin-haptoglobin complex and its levels in an indication of monocyte-macrophage activation. The soluble form of the receptor is called sCD163 and is found in plasma. Plasma sCD163 levels are up-regulated in a large range of inflammatory diseases (16).

Hypothesis Patients with dementia have a deregulated concentration and/or activity of IGF-I, IGF-II, NGF, BDNF and sCD-163 in cerebrospinal fluid.

Purpose To define the concentration and biological activity of IGF-I, IGF-II, BDNF, NGF and sCD-163 in the cerebrospinal fluid and serum in patients with Alzheimer's compared with controls (patients with unspecified neurological symptoms or disease).

Method Study population All participating patients must be over the age of 18 years old. They are excluded from the study in case of acute bacterial neuro infection and acute bleeding The study population of this project will include all patients with established or suspected dementia, who will undergo a lumbar puncture at the Department of Neurology at Aarhus University Hospital as part of their diagnostic work-up.

Controls include patients with unspecified neurological symptoms or diseases who will undergo a lumbar puncture at the Department of Neurology at Aarhus University Hospital as part of their diagnostic work-up irrespective of this study.

The patients will receive information about the research project and will be asked to give their content to participation. The participation implies extraction of 2-3 ml extra of spinal fluid and an extra blood sample(10ml), which will be used for analysis of IGF system components and neurotrophic factors. Participants will not receive any form of payment, but can receive compensation for transportation.

At all times during the diagnostic work-up and consequently in the research project we will take the patients mental and physical condition into consideration. The research project will be carried out according to the Act on Processing of Personal Data.

At the Department of Neurology at Aarhus University Hospital, the Dementia Clinic use lumbar puncture as a diagnostic tool in approximately three patients per week. It is estimated that about 1/3 to 1/2 of these patients will end up with the diagnosis Alzheimer and these patients will ultimately be included in the project during a period of 36-40 weeks. Overall during the study period this will enable inclusion of 50-60 patients.

Analysis The spinal fluid and the serum will be analysed at the Medical Research Laboratory. The spinal fluid and blood samples will be deposited in a research biobank at Aarhus University Hospital. The plan is to carry out all the biochemical analyses at the same time when all samples are collected. In case of knew knowledge in the field we intend to deposit the samples for 5 years after this project. If the samples are to be used for another project The National Committee on Health Research Ethics and the Danish Data Protection Agency will demand an application once more.

The immunological concentrations of IGF-I and IGF-II are measured by validated in-house analyses. Furthermore, Aarhus University Hospital has a unique technique, whereby it is possible to measure the bioactivity of IGF-I and -II in the cerebrospinal fluid. The technique is based on a cell-based in-house bioassay developed in 2003. This method takes in to account that a large part of the IGF-I and IGF-II is bound to proteins and thereby to be considered biological inactive. The bioassay is able to measure the ability of both serum and cerebrospinal fluid to stimulate IGF-IR in vitro which makes the method much more specific. Pilot investigations from our group have shown that it is possible to measure the biological IGF-IR activity in cerebrospinal fluid. It has been proven that:

i) The biological IGF in vitro activity of cerebrospinal fluid primarily comes from IGF-II ii) The biological activity is far higher than expected as compared to simple measures of concentration owing to the low concentrations of IGF-binding proteins.

The immunological concentrations of the IGF-binding proteins will be measured by commercial or in-house developed immunoassays and ligand blotting techniques.

The concentrations of NGF, BDNF and sCD-163 in spinal fluid and serum will be analysed by already established techniques and the spinal fluid will be examined with spectrometry.

Clinical examination The clinical examination will be performed as a natural part of the examination of dementia. This includes medical history and an objective examination, CT scan and cognitive tests including MMSE (mini-mental state examination) and ACE (Adenbrooke´s Cognitive Examination). In the case of doubt a more extended examination will be performed by a neurophysiologist. Information from the clinical examination in form of medical record will be used to evaluate the possibility of dementia as diagnosis including the progression of the disease and thereby to evaluate the possible deregulated concentrations and/or activities of IGF-I, IGF-II, NGF, BDNF and sCD-163 in cerebrospinal fluid.

Power The bioactivity of IGF in cerebrospinal fluid in patients with dementia have not earlier been determined. Pilot data indicate that bioactivity from IGF-II in healthy people(n= 9) is 57 ± 13 ng/ml(mean ± SD). If the difference in a patient group is set to 26ng/ml ( ̴ 2 x SD) then inclusion of 10 persons per group give the project a power of 90% by use of ANOVA and a significant level of 5 %. It has therefore been chosen to include 15 patients in the project.

Statistic The program ANOVA will be used for statistical analyses. Parametric or non-parametric tests will be used depending of the normal distribution of data. In all statistical analysis a 5% level of significance will be used.

Perspective As earlier mentioned the costs of dementia already account for 1% of the world's GDP and the prevalence of dementia is expected to double within the next twenty years. The progressive nature of the disease means that estimated 43% of cases with dementia need a high level of care (equivalent to a nursing home). Therefore, it is obvious that prevention, delayed onset, slowed progression and potential curability are crucial factors for not only the well-being of patients and relatives but also for the economy of the health care systems. (2,17) This research project is based on the recent theory of dementia as a disease in the IGF-system, but as opposed to other studies we are able to measure concentrations as well as bioactivity. This will potentially open up for further knowledge about the dynamic of dementia and thereby potentially reveal further understanding of the pathogenesis and medical targets of dementia.

Ethical consideration Ethical considerations in general The tests performed on the patients involved in this research project are lumbar puncture and blood samples. Both of these tests will be performed as part of the diagnostic workup irrespective of this study.

It involves some risks to perform a lumbar puncture, which include post lumbar puncture headache with a incidence of 12 %, but is most common in younger patients. Most frequently, the headache has a short duration and it may be cured with application of a blood-patch. The use of a needle to the lumbar puncture can cause temporary lumbar pain and an accumulation Ethical considerations for patients with dementia The concerned patient group causes an extended ethical consideration. As mentioned earlier the symptoms of dementia causes memory loss, difficulty in finding the right words and understanding what people are saying. As such it is questionable whether the patients are able to make an independent decision on whether to participate in the project (6).

All of the dementia patients will have all the tests performed as part of the standard diagnostic work up for dementia. Therefore this study does not introduce any additional investigation defending the ethical aspect of this study. In consideration of the low risk involved in this project, the mild dementia forms and the high prevalence and seriousness of the disease we evaluate this project to be ethically acceptable. Furthermore it is of great importance to examine the pathogenesis and possible targets of dementia.

Aim Positive, negative as well as inconclusive results from this study will be published. The results will be the foundation of a research year report and an article for publication in an English written peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* dementia, controls(lumbar puncture at our department)

Exclusion Criteria:

* <18år
* other CNS disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dementia
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Concentration and/or activity of IGF-I in cerebrospinal fluid. | day 1
  People with dementia compared with controls
Concentration and/or activity of IGF-II in cerebrospinal fluid. | day 1
  People with dementia compared with controls
Concentration of NGF in cerebrospinal fluid. | day 1
  People with dementia compared with controls
Concentration of BDNF in cerebrospinal fluid. | day 1
  People with dementia compared with controls
Concentration of sCD163 in cerebrospinal fluid. | day 1
  People with dementia compared with controls

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Aarhus C, Denmark

REFERENCES:
- [Background] Holmes, Clive: Dementia: Medicin(United Kingdom), 2012, Vol. 40, part 11, p. 628-631
- [Background] Georges J, Jansen S, Jackson J, Meyrieux A, Sadowska A, Selmes M. Alzheimer's disease in real life--the dementia carer's survey. Int J Geriatr Psychiatry. 2008 May;23(5):546-51. doi: 10.1002/gps.1984. PMID 18232054
- [Background] Luque FA, Jaffe SL. The molecular and cellular pathogenesis of dementia of the Alzheimer's type an overview. Int Rev Neurobiol. 2009;84:151-65. doi: 10.1016/S0074-7742(09)00408-5. PMID 19501717
- [Background] Bertram L. Alzheimer's disease genetics current status and future perspectives. Int Rev Neurobiol. 2009;84:167-84. doi: 10.1016/S0074-7742(09)00409-7. PMID 19501718
- [Background] Hampel H, Lista S, Teipel SJ, Garaci F, Nistico R, Blennow K, Zetterberg H, Bertram L, Duyckaerts C, Bakardjian H, Drzezga A, Colliot O, Epelbaum S, Broich K, Lehericy S, Brice A, Khachaturian ZS, Aisen PS, Dubois B. Perspective on future role of biological markers in clinical therapy trials of Alzheimer's disease: a long-range point of view beyond 2020. Biochem Pharmacol. 2014 Apr 15;88(4):426-49. doi: 10.1016/j.bcp.2013.11.009. Epub 2013 Nov 22. PMID 24275164
- [Background] Chen DY, Stern SA, Garcia-Osta A, Saunier-Rebori B, Pollonini G, Bambah-Mukku D, Blitzer RD, Alberini CM. A critical role for IGF-II in memory consolidation and enhancement. Nature. 2011 Jan 27;469(7331):491-7. doi: 10.1038/nature09667. PMID 21270887
- [Background] de la Monte SM, Wands JR. Alzheimer's disease is type 3 diabetes-evidence reviewed. J Diabetes Sci Technol. 2008 Nov;2(6):1101-13. doi: 10.1177/193229680800200619. PMID 19885299
- [Background] Hoyer S. Causes and consequences of disturbances of cerebral glucose metabolism in sporadic Alzheimer disease: therapeutic implications. Adv Exp Med Biol. 2004;541:135-52. doi: 10.1007/978-1-4419-8969-7_8. PMID 14977212
- [Background] Bloemer J, Bhattacharya S, Amin R, Suppiramaniam V. Impaired insulin signaling and mechanisms of memory loss. Prog Mol Biol Transl Sci. 2014;121:413-49. doi: 10.1016/B978-0-12-800101-1.00013-2. PMID 24373245
- [Background] Trueba-Saiz A, Cavada C, Fernandez AM, Leon T, Gonzalez DA, Fortea Ormaechea J, Lleo A, Del Ser T, Nunez A, Torres-Aleman I. Loss of serum IGF-I input to the brain as an early biomarker of disease onset in Alzheimer mice. Transl Psychiatry. 2013 Dec 3;3(12):e330. doi: 10.1038/tp.2013.102. PMID 24301648
- [Background] Sopova K, Gatsiou K, Stellos K, Laske C. Dysregulation of neurotrophic and haematopoietic growth factors in Alzheimer's disease: from pathophysiology to novel treatment strategies. Curr Alzheimer Res. 2014 Jan;11(1):27-39. doi: 10.2174/1567205010666131120100743. PMID 24251394
- [Background] Brookmeyer R, Johnson E, Ziegler-Graham K, Arrighi HM. Forecasting the global burden of Alzheimer's disease. Alzheimers Dement. 2007 Jul;3(3):186-91. doi: 10.1016/j.jalz.2007.04.381. PMID 19595937
- See also: About dementia: Alzheimer's disease association — http://www.alz.co.uk/about-dementia